CLINICAL TRIAL: NCT03564379
Title: A Double-blind, Placebo-controlled, Randomized, Single and Multiple Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of JNJ-42165279 in Healthy Japanese Male Subjects
Brief Title: A Single and Multiple Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of JNJ-42165279 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108467; 42165279EDI1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Dose Part (Experimental): Participants will receive a single oral dose of 25 mg JNJ-42165279 or placebo tablet under fasted condition in the morning on Day 1.
  Interventions: Drug: JNJ-42165279; Drug: Placebo
- Part 2: Multiple Dose Part (Experimental): After a washout period of at least 10 days, same participants from Part 1 will receive multiple daily dosing of 25 mg JNJ-42165279 or placebo tablet for 10 days.
  Interventions: Drug: JNJ-42165279; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42165279 — 25 mg JNJ-42165279 tablet will be administered orally.
Drug: Placebo — Matching placebo tablet will be administered orally.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of JNJ-42165279 in healthy Japanese male participants after single and multiple oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of clinical laboratory tests performed at screening and Day -1. If the results of the serum chemistry panel including liver enzymes, other specific tests, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* A man who is sexually active with a woman of childbearing potential, and has not had a vasectomy with confirmation of azoospermia, must agree to use a barrier method of birth control during the study and for 3 months after receiving the last dose of study drug, and his female partner must also use a highly effective form of birth control at least one month prior to the first study dose and continuing until 3 months after the final study dose. Acceptable barrier methods are male condoms with spermicide, and for the female partner a diaphragm or cervical cap with appropriate spermicidal foam, cream, or gel. Highly effective forms of birth control for the female partner are prescribed hormonal implants, contraceptive patches, contraceptive injections, oral contraceptives, and intrauterine device (IUD)
* Body Mass Index (BMI; weight/height^2 [kilogram per meter square {kg/m^2}]) between 18.0 and 30.0 kg/m^2 (inclusive), and body weight not less than 50.0 kilogram (kg)
* Blood pressure (BP) (after the participant is standing for 3 minutes, supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic (orthostatic cut-off, a fall in systolic BP of at least 20 mmHg or diastolic BP of at least 10 mmHg when a person assumes a standing position is exclusionary). If BP is out of range, up to 2 repeated assessments are permitted

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry, coagulation, or urinalysis at screening (and at admission to the study center) as deemed appropriate by the investigator
* Known allergy, hypersensitivity, or intolerance to JNJ-42165279 or its excipients
* Any Grade 2 laboratory toxicity
* History of clinically significant drug and/or food allergies
* History of epilepsy or fits or unexplained black-outs

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Screening up to Day 4
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Day -1 up to approximately 28 days
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 1: Plasma Concentration of JNJ-42165279 | Up to Day 4
  Plasma concentration of JNJ-42165279 will be reported.
Part 2: Plasma Concentration of JNJ-42165279 | Up to Day 14
  Plasma concentration of JNJ-42165279 will be reported.

SECONDARY OUTCOMES:
Part 1: Minimum Observed Fatty Acid Amide Hydrolase (FAAH) Activity in White Blood Cells (WBC) Concentration (Rmin) | Up to Day 4
  Rmin is the minimum observed FAAH activity in WBC concentration during a dosing interval (may or may not be the trough concentration).
Part 2: Minimum Observed FAAH Activity in WBC Concentration (Rmin) | Day 1, Days 10 to 14 and Follow-up (approximately up to 28 days)
  Rmin is the minimum observed FAAH activity in WBC concentration during a dosing interval (may or may not be the trough concentration).
Part 1: Time to Minimum Observed FAAH Activity in WBC Concentration (tmin) | Up to Day 4
  tmin is the time to the minimum observed FAAH activity in WBC concentration occurred during a dosing interval (may or may not be the trough concentration).
Part 2: Time to Minimum Observed FAAH Activity in WBC Concentration (tmin) | Day 1, Days 10 to 14 and Follow-up (approximately up to 28 days)
  tmin is the time to the minimum observed FAAH activity in WBC concentration occurred during a dosing interval (may or may not be the trough concentration).
Part 1: Maximum Percent Change in FAAH Activity in WBCs, Compared to Baseline (Predose) Value of Plasma Fatty Acid Amides (FAA) | Baseline Up to Day 4
  Maximum percent change in FAAH activity in WBCs, compared to baseline (that is, predose) value of Plasma FAA (ethanolamine [AEA], Palmitoylethanolamide/amine [PEA] and Oleoylethanolamide/amine [OEA]) will be observed.
Part 2: Maximum Percent Change in FAAH Activity in WBCs, Compared to Baseline (Predose) Value of Plasma FAA | Baseline, Day 1, Days 10 to 14 and Follow-up (approximately up to 28 days)
  Maximum percent change in FAAH activity in WBCs, compared to baseline (that is, predose) value of Plasma FAA (AEA, PEA, and OEA) will be observed.
Part 1: Plasma Concentrations of Fatty Acid Amides (FAAs - N-Arachidonoyl ethanolamine [AEA], Palmitoylethanolamide/amine [PEA] and Oleoylethanolamide/amine [OEA]) | Up to Day 3
  Plasma concentration of FAAs including AEA, PEA, and OEA will be reported.
Part 2: Plasma Concentrations of FAAs (AEA, PEA and OEA) | Day 1 and Days 10 to 14
  Plasma concentration of FAAs including AEA, PEA, and OEA will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- WCCT Global, LLC, Cypress, California, United States